CLINICAL TRIAL: NCT01268904
Title: Safety and Efficacy of Intravenous Valproate in Pediatric Status Epilepticus and Acute Repetitive Seizures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Iyad Magadly, Hillel Yaffe Medical Center
Other Study IDs: 0098-10-HYMC
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Valproic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pediatric status epilepticus
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate — Intravenous valproate application to pediatric patients suffering from status epilepticus and acute repetitive seizures

SUMMARY:
To evaluate the safety and efficacy of intravenous valproate in pediatric status epilepticus and acute repetitive seizures as part of seizure treatment protocol in pediatric ER

ELIGIBILITY:
Inclusion Criteria:

* Child with clinical presentation of status epilepticus

Exclusion Criteria:

* All others

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric inpatients and emergency patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Safety of intravenous valproate in pediatric status epilepticus | One week

SECONDARY OUTCOMES:
Efficacy of intravenous valproate in pediatric status epilepticus | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel